CLINICAL TRIAL: NCT00597194
Title: Day Case Inguinal Hernia Repair in Children. Is Laparoscopic Approach Justified?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Children and Adolescents, Finland (Other)
Responsible Party: Professor Christer Holmberg, Hospital for Children and Adolescents, Helsinki, Finland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 216L2002; T 1040L0007
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2007-12

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; laparoscopic repair; open repair; randomized
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OH (Active Comparator): Inguinal hernia operated using a classic open herniotomy(OH)
  Interventions: Procedure: Hernia repair
- LH (Active Comparator): Laparoscopic herniorraphy (LH) for inguinal hernia
  Interventions: Procedure: Hernia repair

INTERVENTIONS:
Procedure: Hernia repair — Hernia repair laparoscopically (LH) or by open operation (OH)

SUMMARY:
We compare laparoscopic and classic open operation for inguinal hernia in children. Attention is focused on the recovery, surgical result and the duration of the operation and hospital stay.

DETAILED DESCRIPTION:
Background and objective : In adults the advantages laparoscopic inguinal hernia are less pain, shorter recovery, shorter sick leave and better cosmetic result. It is not known whether laparoscopic hernia repair produces similar results in children.The objective is to compare the duration of recovery, postoperative pain and long-term surgical results between day case laparoscopic and open inguinal hernia repair in children.

Key inclusion criteria: Children included in the study must be aged four months to sixteen years of age and not have undergone any previous surgery. Of male patients those with completely descended testes are accepted.

Study type: The study is randomized, single-blinded prospective comparison between laparoscopic and open day case inguinal hernia repair in children.

Target sample size: For the assumption that there is a difference of one day in time to restore normal activities after laparoscopic and open hernia repair, target sample size of 100 patients in the laparoscopic and 100 in open repair arm should reach 90% power with p < 0.05.

Recruitment status : From 10/ 2002 to 1/2007 89 patients (laparoscopic repair LH 47, open repair OH 42) are recruited. Primary outcome: The time to restore normal activity after surgery . Secondary Outcomes : The degree of postoperative pain, the duration of the operation, sick leave of parents, surgical result 6 months and 2 years after the repair.

ELIGIBILITY:
Inclusion Criteria:

* unilateral inguinal hernia
* age age > 4 months, <16 years
* fully descended testes
* study consent signed

Exclusion Criteria:

* previous abdominal or inguinal surgery
* testes not fully descended
* not healthy enough for day surgery
* age < 4months or >16 years
* study consent not signed

Ages: 4 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2002-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
recovery after inguinal hernia surgery = time to restore normal activities after surgery | one week

SECONDARY OUTCOMES:
degree of postoperative pain | 3 days
duration of surgery and hospital stay | 1 day
long term surgical result | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Antti I Koivusalo, MDPhD, Principal Investigator — Hospital for Children and Adolescents,Helsinki,Finland; Mikko P Pakarinen, MD PhD, Principal Investigator — Hospital for Children and Adolescents,Helsinki,Finland; Risto J Rintala, Professor, Principal Investigator — Hospital for Children and Adolescents,Helsinki,Finland; Christer Holmberg, Professor, Study Director — Hospital for Children and Adolescents,Helsinki,Finland
Locations (1):
- Hospital for Children and Adolescents, Helsinki, Finland

REFERENCES:
- [Background] Butler RE, Burke R, Schneider JJ, Brar H, Lucha PA Jr. The economic impact of laparoscopic inguinal hernia repair: results of a double-blinded, prospective, randomized trial. Surg Endosc. 2007 Mar;21(3):387-90. doi: 10.1007/s00464-006-9123-6. Epub 2007 Jan 19. PMID 17235721
- [Background] Eklund A, Rudberg C, Smedberg S, Enander LK, Leijonmarck CE, Osterberg J, Montgomery A. Short-term results of a randomized clinical trial comparing Lichtenstein open repair with totally extraperitoneal laparoscopic inguinal hernia repair. Br J Surg. 2006 Sep;93(9):1060-8. doi: 10.1002/bjs.5405. PMID 16862612
- [Background] Schier F. Laparoscopic inguinal hernia repair-a prospective personal series of 542 children. J Pediatr Surg. 2006 Jun;41(6):1081-4. doi: 10.1016/j.jpedsurg.2006.02.028. PMID 16769338
- [Derived] Koivusalo AI, Korpela R, Wirtavuori K, Piiparinen S, Rintala RJ, Pakarinen MP. A single-blinded, randomized comparison of laparoscopic versus open hernia repair in children. Pediatrics. 2009 Jan;123(1):332-7. doi: 10.1542/peds.2007-3752. PMID 19117900